CLINICAL TRIAL: NCT04381988
Title: A Phase II Randomized Double-Blind Placebo-Controlled Clinical Trial Of Hydroxychloroquine For Prophylaxis Against Covid-19 In Patients Receiving Radiotherapy (COVID)
Brief Title: A Study of Hydroxychloroquine vs Placebo to Prevent COVID-19 Infection in Patients Receiving Radiotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated based results of other studies and use of the new vaccine.
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20-176
Record Dates: First submitted 2020-05-08; First posted 2020-05-11 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-04

CONDITIONS: COVID-19; Cancer
Keywords: Hydroxychloroquine; Radiotherapy; 20-176
MeSH Terms: conditions — COVID-19; Neoplasms | interventions — Hydroxychloroquine; Radiotherapy

STUDY DESIGN:
Intervention Model Description: This is a randomized (1:1), double-blind, placebo-controlled phase II clinical trial.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Experimental): Every patient on trial must be scheduled to receive at least 10 radiation treatments prior to initiation of hydroxychloroquine 400mg daily.
  Interventions: Drug: Hydroxychloroquine; Radiation: Radiation therapy
- Placebo (Placebo Comparator): Every patient on trial must be scheduled to receive at least 10 radiation treatments prior to initiation of placebo 400mg daily.
  Interventions: Other: Placebo; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Hydroxychloroquine — 400mg daily
  Arms: Hydroxychloroquine
Other: Placebo — 400mg daily
  Arms: Placebo
Radiation: Radiation therapy — Standard radiation therapy will be prescribed and administered as per the patient's radiation oncologist.

SUMMARY:
The researchers are doing this study to find out whether the study drug hydroxychloroquine can prevent infection with the COVID-19 virus, compared with placebo, in people who are receiving radiation therapy for their cancer. The placebo used in this study is a tablet that looks the same as the study drug and is taken in the same way, but it does not contain any active ingredients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* ECOG 0-3
* For patients who have not started radiation at the time of screening: patients are required to have a plan in place for a minimum of 10 radiation treatments with or without concurrent systemic therapy
* For patients who have already started radiation at the time of screening: patients must complete enrollment such that they are able to receive at least 10 radiation treatments with hydroxychloroquine.
* Disease Site
* Mandatory inclusion criteria:
* No COVID-19 symptoms within 14 days of enrollment:

  * (Temp >38C in addition to sore throat, cough, wheezing, chest tightness, shortness of breath, body aches, chills, diarrhea, and anosmia)
  * If symptoms are present within 14 days of enrollment, patients with a negative COVID-19 PCR or COVID-19 serology assay are eligible for inclusion.
* No close contact with confirmed COVID-19 person
* Close contact defined as:

  * Within 6 feet for prolonged period
  * Cohabitating
* Optional laboratory criteria (Recommended if available)

  * Negative pre-treatment SARS-CoV-2 rapid antigen test result (within 1 week of enrollment)
  * Negative pre-treatment SARS-CoV-2 PCR test result (within 1 week of enrollment) using MSKCC laboratory or outside laboratory assay
  * Negative pre-treatment Standard Q COVID-19 IgM/IgG rapid serology result (within 1 week of enrollment)
  * Blood serum for SARS-CoV-2 serology tests (being validated by MSKCC)
* Disease site meets following criteria:

  * Head and Neck / High-Risk Skin Cancer
  * Lung Cancer
  * Breast Cancer
  * Prostate Cancer
  * Central Nervous System Tumors
  * Gastrointestinal System Cancer
  * Gynecologic cancer
  * Other disease sites permitted at PI discretion

Exclusion Criteria:

* Previous positive test for SARS-CoV-2
* Previous positive serology test for SARS-CoV-2
* Recent Chest CT meeting CT exclusion criteria
* Live in a skilled nursing facility with COVID-19 symptoms (Temp >38 C in addition to sore throat, cough, wheezing, chest tightness, shortness of breath, body aches or chills, diarrhea, anosmia)
* Known hypersensitivity to hydroxychloroquine or 4-aminoquinoline derivatives
* Pre-existing retinopathy
* Known chronic kidney disease, stage 4 or 5, or receiving dialysis
* Breast Feeding
* Tamoxifen
* Absolute neutrophil Count <1,000/ml at registration
* Concurrent use of any other quinine derivative
* Antiarrhythmic medications: amiodarone, sotalol, dofetilide, procainamide, quinidine, flecainide
* Glucose-6-phosphate dehydrogenase deficiency
* Pre-treatment corrected QT interval (QTc) ≥470 milliseconds**
* Prisoners
* Inability to participate
* Psoriasis
* History of suicidal ideation
* CT Criteria for Enrollment Exclusion (Optional - only for patients who received a diagnostic CT as part of standard of care or a thoracic CT as part of radiation simulation): All patients with COVID-19 typical radiographic findings on CT Chest as defined by the RSNA will be excluded. Patients with any NEW COVID-19 indeterminate radiographic findings on CT Chest that are concerning for COVID-19 will be excluded. COVID-19 indeterminate features are permitted if they can be demonstrated as STABLE on prior (>14 calendar days) CT Chest or PET/CT. If no prior comparison is available AND any intermediate or typical feature is present, the patient is not eligible.
* COVID-19 Atypical Features

  * Isolated lobar or segmental consolidation without GGO
  * Discrete small nodules (centrilobular, "tree-in-bud")
  * Lung cavitation
  * Smooth interlobular septal thickening with pleural effusion
* COVID-19 Indeterminate Features

  * Multifocal, diffuse, perihilar, or unilateral GGO with or without consolidation lacking a specific distribution and are non-rounded or non-peripheral
  * Few very small GGO with a non-rounded and non-peripheral distribution
* COVID-19 Typical Features

  * Peripheral, bilateral GGO with or without consolidation or visible intralobular lines ("crazy paving")
  * Multifocal GGO of rounded morphology with or without consolidation or visible intralobular lines ("crazy paving")
  * Reverse Halo sign or other findings of organizing pneumonia ** If pre-treatment QTC can be decreased to <470, the patient can be re-considered for trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memoral Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memoral Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All Protocol Activities), Commack, New York
  - Memoral Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydroxychloroquine | Placebo
Started | 4 | 0
Completed | 0 | 0
Not Completed | 4 | 0
Not completed — The study was terminated | 4 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated before more participants were accrued.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine | Placebo | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Continuous [Mean (Full Range); unit: years] | 63 [58 to 70] |  | 63 [58 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 0 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of SARS-CoV-2 Infection
Description: Any patients who are enrolled and subsequently test positive for SARS-CoV-2 by RT-PCR (outside RT-PCR test results allowed) at any point during the 9 weeks following enrollment will be an event that is considered in the 9-week SARS-CoV-2 infection rate primary endpoint.
Time Frame: within 9 weeks from randomization
Population: Data were not collected.
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Cumulative Incidence of Severe COVID-19 or Death
Description: Patients who are positive for SARS-CoV-2 (as defined above) who develop a new oxygen requirement attributable to COVID-19, tachypnea (RR > 20), or those who require hospitalization due to COVID-19 will be considered to have severe COVID-19.
Time Frame: within 12 weeks of randomization
Population: Data were not collected
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: The study was terminated based results of other studies and use of the new vaccine
Arm/Group | Hydroxychloroquine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 0/4 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT04381988/Prot_SAP_000.pdf